CLINICAL TRIAL: NCT04927221
Title: A Randomized, Double-Blind, Placebo-Controlled Phase Ib/IIa Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of DC739 Multiple-Dose in Hypercholesterolemic Subjects.
Brief Title: Multiple Ascending Dose Study to Evaluate the Safety, Tolerability of DC371739 Treatment in Hypercholesterolemic
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou JOYO Pharma Co., Ltd (Industry)
Collaborators: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JYD0102
Record Dates: First submitted 2021-05-29; First posted 2021-06-15 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2021-05

CONDITIONS: Hypercholesterolemia
Keywords: Hypercholesterolemia; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of 5 groups in parallel for the duration of the study
Who Masked: Participant
Masking Description: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DC371739 20mg Dose MAD (Experimental): Orally administered DC371739 tablets QD afer meal
  Interventions: Drug: DC371739 Tablets
- DC371739 Placebo MAD (Placebo Comparator): Placebo orally administered
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DC371739 Tablets — Participants received one of 5 dose levels of DC371739 administered as single oral doses.
  Arms: DC371739 20mg Dose MAD
Drug: Placebo — Placebo orally administered as comparison
  Arms: DC371739 Placebo MAD

SUMMARY:
This study is to evaluate safety, tolerability, pharmacokinetics and pharmacodynamics of DC739 after multiple-dose oral administration, to explore the clinical effective dose, and to initially explore the efficacy and safety in hypercholesterolemia subjects.

DETAILED DESCRIPTION:
Totally about 30-50 qualified subjects were assigned to one of the following dose groups：20mg, 40mg, 60mg, 80mg, 120 mg (60mg and 120mg is the optional dose group). Each of the dose groups will include 10 subjects (8 for DC739 and 2 for placebo).

Subjects will be admitted for treatment on day -1 and receive the first dose of study drug or placebo on day 1 and then treat for 28 days. Subjects from different dose groups were enrolled in turn, the next dose group is conducted on the premise that the D15 safety evaluation was completed after the administration of the previous dose group with the result was tolerance.

Blood samples will be collected on day 1 for 48 hours and day 28 for 72 hours after administration for pharmacokinetic data analysis. Blood lipid will be collected for effectiveness evaluation. PCSK9 and ANGPTL3, Urine and feces were collected for explore analysis.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 65 years (inclusive 18 and 65);
* Body mass index of 18 to 32 kg/m2(inclusive);
* Hypercholesterolemia subjects with LDL-C≥2.6mmol/L(100mg/dL);
* Male or female subjects who had no immediate plans to have children, the serum pregnancy test of women was negative at the time of screening, and agreed to use strict contraceptive measures throughout the study period and up to 6 months after the last dose;

Exclusion Criteria:

* ECG confirmed that the QT interval was prolonged > 450ms (QT interval corrected for heart rate by Bazetts formula [QTCB]);
* Use of statins (lovastatin, simvastatin, pravastatin, mevastatin, fluvastatin, atorvastatin, cerivastatin, rosuvastatin, pitavastatin, etc.) , ezetimibe, Xuezhikan, and other lipid-lowering treatment within 2 months prior to screening; use of PCSK9 monoclonal antibodies , fibric acid drugs (such as fenofibrate, gemfibrozil) and probucol within 3 months prior to screening;
* Use of warfarin, systemic steroids, cyclosporine, or other immunosuppressive therapy within months prior to screening;
* Subjects with HIV-AB , HBsAg, ANTI-TP , HCV-AB positive;
* A history of prescription drug abuse and illicit drug abuse within 6 months prior to screening;
* A history of alcohol abuse within 6 months prior to screening;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
tolerability evaluation | From informed consent until Day 42.
  12-lead ECG
Safety evaluation | From informed consent until Day 42.
  adverse events (AE/SAEs)
Pharmacodynamic evaluation | From informed consent until Day 31.
  Cmax

SECONDARY OUTCOMES:
Effective evaluation | From informed consent until Day 29.
  LDL-C

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Derived] Wang J, Zhao J, Yan C, Xi C, Wu C, Zhao J, Li F, Ding Y, Zhang R, Qi S, Li X, Liu C, Hou W, Chen H, Wang Y, Wu D, Chen K, Jiang H, Huang H, Liu H. Identification and evaluation of a lipid-lowering small compound in preclinical models and in a Phase I trial. Cell Metab. 2022 May 3;34(5):667-680.e6. doi: 10.1016/j.cmet.2022.03.006. Epub 2022 Apr 14. PMID 35427476